CLINICAL TRIAL: NCT06046651
Title: Blood Specimen Collection For Laboratory Assay Research
Status: Recruiting | Type: Observational
Sponsor: Roman Health Ventures Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RS.0723.012
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: General; Metabolic Disorder; Sexual Dysfunction; Hair Loss; Pathology
MeSH Terms: conditions — Metabolic Diseases; Sexual Dysfunction, Physiological; Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To collect lab data from capillary and venous blood specimens for use in analytical research studies to support the development and validation of laboratory procedures.

DETAILED DESCRIPTION:
Introduction Overview Remote health monitoring is becoming more commonplace in traditional and non-traditional medical practices, including for the analysis of blood. As venipuncture processes may cause distress and lead to lower patient compliance, the ability to collect blood through capillary samples is becoming increasingly popular due to patient demand and the limited availability of phlebotomists. With recent advances in lab instrumentation, the ability to analyze small volumes of blood to support the diagnostic process is gradually becoming more established.

Despite the development of several novel devices to collect capillary samples, limited data is available on the stability of such samples across various environmental conditions and lengths of time. In addition, there continues to be a need to compare the correlation between lab results obtained from capillary samples, as compared to venous samples, which is the gold standard. The aim of this study is to collect capillary (fingerstick) blood samples and under various circumstances, assess their viability for broad-based consumer lab testing.

Background Traditionally, clinical lab results have been limited to data collected from select sites that have phlebotomists on-site. While valuable, these diagnostic services are only available to individuals who live close enough to a lab, thereby limiting our understanding of disease within the broader community. Lab visits are limited to very specific episodes of care, which exclude the ability to remotely monitor the progression of disease. In addition, these limited lab visits usually only study a small set of assays within each individual, biasing our understanding of any other underlying medical conditions that exist within a population. The need to develop technology to make diagnostic services more accessible is paramount to not only better treat acute and chronic diseases, but to also support behavioral change toward the prevention of disease.

At-home blood collection for lab testing has become increasingly popular to monitor disease and access treatments more rapidly. The ability to broaden access to diagnostic testing, especially in healthcare deserts, is valuable to mitigating the progression of disease. For example, clinicians will have access to a higher volume of lab data and be able to identify disease patterns more readily, which may lead to quicker intervention. On a population health level, improved access to diagnostics will provide insights into patient behavior and underlying disease states that may otherwise not be observed.

Empowering patients to collect their own samples will provide a longitudinal view of disease, and enable deeper discussions with their clinicians regarding appropriate treatment and lifestyle changes.

Study Design This is an internal observational study, non-interventional.

Methods Sample Collection and Handling Specimens will either be self-collected by the subject (capillary samples) or collected by a licensed healthcare professional (capillary or venous samples) at the investigator's wholly-owned facility or a subject's home. Specimens will be stored or transported to one of the investigator's laboratories, a third-party laboratory, or a research facility for use in analytical research studies.

Subjects may elect to provide a single sample, or continue providing samples on a regular basis until the subject withdraws from the study, is removed from the study, or the study is closed. Study visits are limited to 1 visit per 24 hour period.

Specimen Type and Collection Methods Specimen Collection Method Capillary Blood Capillary blood will be collected from a finger using a standard lancet, by the subject independently or with the assistance of a licensed healthcare professional.

Collection instructions, following consent:

Either independently, or under the direction of research staff, apply a hand warmer on the desired finger or run the finger under warm water for 1 minute. Dry finger. Clean skin with an alcohol wipe, and allow the alcohol to dry. Apply lancet to finger. Drip blood into a specified collection container, which may be a capillary tube or other blood transfer device. Notwithstanding any other specimen collections described in this protocol, a maximum of 4 capillary blood draws may be collected in one visit (less than 4 mL total).

At-home kit:

When subjects collect their own samples off-site, all necessary containers, materials, and instructions for shipping will be included in the original collection kit. Shipment will be designed to comply with packaging associated with "Exempt human specimen."

Shipment preparation procedure will be as follows: Sample is placed in a sealed primary receptacle (tube, vial, container), then secondary packaging (cushioning and absorbent materials), and then into outer packaging.

Venous Blood Venous blood will be collected from the antecubital fossa, forearm, or hand of the subject by a licensed health professional: phlebotomist, physician, nurse, or physician assistant. This collection may occur on-site at the investigator's facility, the subject's home or office, or at any location that is appropriate and convenient.

Collection instructions, following consent:

The investigators will obtain consent from the subject and schedule the subject for phlebotomy at a specific time and site. The healthcare professional performing the specimen collection will confirm with the subject that the subject has provided consent, and confirms that the subject understands that the blood collection will be for research purposes, including for commercial product development, and not for the purpose of diagnosis or treatment. The subject's name and date of birth will be confirmed by the healthcare professional. Additional personal health and demographic information may be collected at this time or any other time during the visit.

Venipuncture: The arm will be prepared with a tourniquet and disinfected with an alcohol pad. Up to 5 tubes (approximately 25 mL) of blood may be collected. After the application of sterile gauze, the needle will then be removed and pressure maintained for at least 1 minute. Following visual examination for any side effects, the venipuncture site will be dressed with a bandage on top of the gauze to apply mild pressure to the venipuncture site. Alternatively, pressure will be maintained for at least 3 minutes with gauze, followed by the application of a self-adhesive bandage.

Sample Processing Blood specimens collected under this protocol will be processed to assess specific study endpoints intended to support the development and validation of laboratory assays and procedures.

Variables of interest may include but are not limited to Temperature Variations: The aliquots may be subjected to different temperature ranges representative of real-life situations, such as refrigerated (2-8°C), room temperature (20-25°C), and elevated temperatures (e.g., > 37°C). Some stability studies might also include extreme temperatures to assess how the sample performs under stress conditions.

Time Points: Each aliquot may be assessed at multiple time points to evaluate the stability of the specimen over time. Common time points for stability testing could be 0 hours (baseline), 24 hours, 48 hours, 72 hours, and so on, depending on research objectives.

Component Separation: Depending on the type of research being conducted, the blood specimens may undergo component separation. This process involves centrifugation to separate the different blood components - plasma, serum, and cellular elements (red and white blood cells). This separation allows the individual components to be analyzed independently, providing valuable insights into how each component behaves during research.

Humidity: Assessing the impact of varying levels of humidity on blood specimen stability, especially in climates with high moisture content.

Light Exposure: Investigating how exposure to different light conditions (e.g., natural light, fluorescent light) might influence the stability of certain analytes in the blood.

Freeze-Thaw Cycles: Replicating scenarios where specimens experience repeated freezing and thawing to evaluate the effects on sample integrity.

Anticoagulants and Additives: Exploring the impact of different anticoagulants or additives on specimen stability to optimize blood collection tubes and preservation methods.

Shipping and Transportation Conditions: Studying the stability of blood specimens during transit and evaluating the impact of varying transportation conditions.

Specimen Volume: Investigating whether different specimen volumes influence stability and testing accuracy.

Freezer or Fridge Storage: Examining the stability of blood specimens under long-term refrigerated or freeze storage conditions (e.g., -20°C, -80°C).

pH and Buffering Conditions: Assessing the role of pH and buffering systems in maintaining the stability of blood components.

Hemolysis and Clot Formation: Investigating the impact of hemolysis and clot formation on test results and evaluating their effects on specimen stability.

The list of variables mentioned above is not exhaustive, and additional factors may be considered based on the specific objectives of the research study.

Procedure Screening / Consent Potential subjects will complete screening using an electronic form, including a brief medical history. Potential subjects will undergo informed consent.

Sample Collection Subjects will attend the study visit at the clinic to have blood samples collected OR Subjects will self-collect samples at home following provided instructions and ship samples to the designated laboratory.

Upon completion of sample collection, subjects will be compensated for their participation and dismissed from the study visit. Subjects may choose to remain enrolled in the study and participate in future study visits, or withdraw from study participation at any time.

Potential Risks and Benefits This research falls under a minimal risk category. The probability of harm or discomfort is comparable to routine clinical examination. All specimen collection is routine with minimal risk of persistent bleeding or infection. There are no direct benefits to the subjects. Research performed based on the collected samples may lead to advances in medical research and commercial (for-profit) products with societal benefits.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, in good general health
* Must be 18 years old or older, inclusive at enrollment
* Must be willing to provide capillary blood samples via a fingerstick and venous blood samples, including self-collection and collection by a licensed healthcare professional
* Must be able to read, understand, and willingly sign an Informed Consent Form (ICF) and complete a brief health questionnaire
* Must be able to read, speak and understand English
* Must be available to attend one study visit at Investigator's laboratory or a third-party laboratory designated by the Investigator or collect samples at home, at the discretion of the Investigator.

Exclusion Criteria:

* Individuals who are unable to provide a blood sample due to any illness
* Individuals participating in another research study, that the Investigator feels may compromise study outcomes
* Individuals having an acute or chronic disease or medical condition, including pregnancy, which could excessively increase study risk in the opinion of the Investigator or compromise study outcomes
* Individuals who are unlikely to be available for the duration of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy members of the community aged 18 years and over
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2033-07-31 (Estimated); Study Completion 2033-08-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between capillary and venous samples upon collection | 10 years
  R-value comparing the lab readings generated by venous and capillary samples for a specific blood analyte immediately upon collection
Stability of the capillary blood sample after storage on Days 1, 2, and 3 | 10 years
  Median error % to compare the difference in values of each capillary sample after storage for a certain period of time (e.g., Days 1, 2, and 3) for a specific analyte when compared to the lab reading generated by the venous sample immediately upon collection

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Vaswani, MD, Principal Investigator — Principal Investigator
Locations (1):
- Roman Health Ventures Study Site, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers